CLINICAL TRIAL: NCT02860078
Title: Comparative Study of the Use of Ultrasonography (USG) or Isolated Use of Fluoroscopy for Sacral Epidural Puncture Corticosteroid Infiltration in Patients With Low Back Pain by Canal Stenosis Lumbar
Brief Title: Epidural Injection of Corticosteroids Under USG (EICUS)
Acronym: EICUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient drug supply
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, SHIRLEY ANDRADE SANTOS, M.D., University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 56795916.8.0000.0068
Record Dates: First submitted 2016-07-17; First posted 2016-08-09 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Pain Management
Keywords: pain; epidural; ultrasound
MeSH Terms: conditions — Agnosia; Pain | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Active Comparator): The group I will be subjected to epidural infiltration using methylprednisolone acetate diluted in ropivacaine 0.1%. Initially the sacral hiatus is identified by palpation. After, the ultrasound device is used (USG) for the puncture, with a linear transducer of high frequency. At the end of corticosteroid administration, the placement of the needle tip will be checked with fluoroscopy and noted.
  Interventions: Device: Ultrasound
- Radioscopy (Active Comparator): The group II will be subjected to infiltration using methylprednisolone acetate diluted in ropivacaine 0.1% . However, only radioscopy be used to guide the puncture.
  Interventions: Device: Radioscopy

INTERVENTIONS:
Device: Ultrasound — Location and function of sacral epidural space with ultrasound
  Arms: Ultrasound
Device: Radioscopy — Location and puncture of the sacral epidural space only with fluoroscopy
  Arms: Radioscopy

SUMMARY:
Qualitative and quantitatively evaluate the pain control and incidence of adverse effects in patients undergoing corticosteroid infiltration and local anesthetic through sacral epidural puncture with ultrasound assistance or isolated use of fluoroscopy to aid puncture and location of the sacral epidural space. A group will be submitted to epidural corticosteroid infiltration associated with local anesthetic with the use of fluoroscopy for locating the sacral epidural space, which is currently the gold standard for this technique, while in another location group will be held with the use of ultrasound.

DETAILED DESCRIPTION:
Introduction: Procedures guided by ultrasound (USG) have advantages over traditional techniques (fluoroscopy) with respect to regional anesthesia. Some studies have shown its usefulness as a quick, safe and simple tool for the location of the sacral hiatus and to guide the puncture of the sacral epidural space in patients with chronic low back pain, despite the lack of data with respect to clinical outcomes.

OBJECTIVES: Evaluate qualitatively and quantitatively the pain control and incidence of adverse effects in patients undergoing corticosteroid infiltration and local anesthetic through sacral epidural puncture with ultrasound assistance or isolated use of fluoroscopy to aid puncture and location of the sacral epidural space. It will also be evaluated success rate in the first puncture, and the time duration of the procedure in groups.

METHODS: It is clinical, analytical, prospective trial, randomized, covered for evaluators. It will include 30 patients with chronic low back pain or pain in the lower limbs resulting in lumbar canal stenosis, refractory to medical treatment. A group will be submitted to epidural corticosteroid infiltration associated with local anesthetic with the use of fluoroscopy for locating the sacral epidural space, which is currently the gold standard for this technique, while in another location group will be held with the use of ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old;
* Patients who have low back and/or lower extremities due to lumbar spinal stenosis pain outpatients, with regular follow-up refractory to conservative medical treatment (Verbal Scale of Pain > 3, more three months duration, with no improvement with clinical treatment).

Exclusion Criteria:

* Symptoms that characterize a surgical emergency;
* The presence of sensory or motor deficit (chronic mild motor impairment or mild paresthesia will not be deleted), injury to peripheral nerves, trauma history or recent fracture;
* Serious medical conditions or decompensated;
* Infection at the puncture site;
* Coagulopathy;
* Contrast allergy history or the medications used in the technique;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-01-17 (Actual)

PRIMARY OUTCOMES:
Pain management | 1 year
  After infiltration, the patient will be reassessed as to pain control in 15 days, 3, 6 and 12 months. Pain is assessed using a verbal analog scale (VAS) from 0 to 10, with 0 being no pain and 10 being the worst possible pain. Patients will quantify the pain at rest, improvement factors and worse, smaller and higher scores during the day, and average daily pain.
Satisfaction with treatment | during the procedure
  Satisfaction with the treatment of pain is assessed using a numerical scale from 0 to 10, 0 being unsatisfied and 10 being complete satisfaction.
Medications | 3 months
  It will be noted and all medications used by the patient before the procedure, and their doses, repeating the notes after 3 months of follow-up after the block.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Andrade Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chen CP, Tang SF, Hsu TC, Tsai WC, Liu HP, Chen MJ, Date E, Lew HL. Ultrasound guidance in caudal epidural needle placement. Anesthesiology. 2004 Jul;101(1):181-4. doi: 10.1097/00000542-200407000-00028. PMID 15220789
- [Result] Marhofer P, Schrogendorfer K, Koinig H, Kapral S, Weinstabl C, Mayer N. Ultrasonographic guidance improves sensory block and onset time of three-in-one blocks. Anesth Analg. 1997 Oct;85(4):854-7. doi: 10.1097/00000539-199710000-00026. PMID 9322469
- [Result] Marhofer P, Schrogendorfer K, Wallner T, Koinig H, Mayer N, Kapral S. Ultrasonographic guidance reduces the amount of local anesthetic for 3-in-1 blocks. Reg Anesth Pain Med. 1998 Nov-Dec;23(6):584-8. doi: 10.1016/s1098-7339(98)90086-4. PMID 9840855
- [Result] Manchikanti L, Knezevic NN, Boswell MV, Kaye AD, Hirsch JA. Epidural Injections for Lumbar Radiculopathy and Spinal Stenosis: A Comparative Systematic Review and Meta-Analysis. Pain Physician. 2016 Mar;19(3):E365-410. PMID 27008296
- [Result] Manchikanti L, Singh V, Cash KA, Pampati V, Damron KS, Boswell MV. Effect of fluoroscopically guided caudal epidural steroid or local anesthetic injections in the treatment of lumbar disc herniation and radiculitis: a randomized, controlled, double blind trial with a two-year follow-up. Pain Physician. 2012 Jul-Aug;15(4):273-86. PMID 22828681
- [Result] Blanchais A, Le Goff B, Guillot P, Berthelot JM, Glemarec J, Maugars Y. Feasibility and safety of ultrasound-guided caudal epidural glucocorticoid injections. Joint Bone Spine. 2010 Oct;77(5):440-4. doi: 10.1016/j.jbspin.2010.04.016. Epub 2010 Sep 24. PMID 20869897